CLINICAL TRIAL: NCT05852080
Title: Multilevel System Intervention Based on Information Platform to Reduce Stroke Recurrence Rate in Acute Ischemic Stroke Patients
Brief Title: Multilevel System Intervention Based on Information Platform to Reduce Ischemic Stroke Recurrence Rate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MISA
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-04

CONDITIONS: Acute Ischemic Stroke; Stroke Recrudescence; Quality Improvement
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm (Experimental): Hospitals in the intervention arm will receive a multilevel system intervention based on information platform
  Interventions: Behavioral: multilevel system intervention based on information platform
- control arm (No Intervention): Hospitals in the control arm will receive no intervention

INTERVENTIONS:
Behavioral: multilevel system intervention based on information platform — 1. Standardized templates of medical record
  2. Continuous medical quality control and feedback system: the hospital included in the study upload the medical records of all AIS patients by medical records scanning system. Quality control platform of Cerebral apoplexy in Zhejiang province extracts and analyze the data through the computer and calculates the percentage of stroke of undetermined cause.
  3. Team collaboration based on video conferencing: hospitals will receive corresponding suggestions for their improvement from experts online.
  4. Enhanced feedback incentives
  Arms: intervention arm

SUMMARY:
A prospective, multicenter and cluster randomised controlled trial will be conducted, using hospital as randomisation unit. Hospitals in Zhejiang Province, China, will be randomised into two arms (1:1): an intervention arm and a control arm. Hospitals in the intervention arm will receive a multilevel system intervention based on information platform, whereas hospitals in the control arm will receive no intervention. The randomisation will be conducted after baseline data collection. The following baseline data will be used for randomisation match: hospital classification, beds in stroke centre, and the number of acute ischemic stroke (AIS) patients within 7 days of stroke onset. Hospitals with <250 AIS cases per year will be excluded from the study. The primary outcome will be difference between intervention arm and control arm in the one-year stroke recurrence rate on the follow-up stage (post-intervention).

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 years or older.
* Patients admitted with neurological deficit consistent with ischemic stroke within 7 days of of symptoms onset. (*Symptom onset is defined by the "last seen normal" principle)
* Confirmation of new ischemic stroke by objective modality of CT scan and MRI (had relevant lesions on DWI).
* Informed consent from patient or legally authorised representative (primarily spouse, parents, adult children, otherwise indicated).

Exclusion Criteria:

* Patients refuse to participate in this study.
* Patients who losing his medical record of having the incomplete medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of new ischemic stroke events | 1 year
  To evaluate the efficacy of intervention in reducing the risk of new ischemic stroke events at 1 year after initial symptom onset.

SECONDARY OUTCOMES:
Incidence rate of new ischemic stroke events | 3, 5 years
  Incidence rate of new ischemic stroke events at 3, 5 years after initial symptom onset.
Incidence rate of new clinical vascular events (ischemic stroke, hemorrhagic stroke, myocardial infarction) | 1, 3, 5 years
  incidence rate of new clinical vascular events (ischemic stroke, hemorrhagic stroke, myocardial infarction) at 1, 3, 5 years after initial symptom onset.
All-cause mortality | 1, 3, 5 years
  All-cause mortality
The percentage of stroke of undetermined cause at discharge | 1 year
  The percentage of stroke of undetermined cause at discharge
Rate of antithrombotic therapy at discharge | 1 year
  The rate of patients with cerebral infarction who received antithrombotic drugs (such as aspirin, other antiplatelet agents, heparin, warfarin or new oral anticoagulants) at discharge in the total number of hospitalized patients with cerebral infarction in the same period.
Rate of anticoagulant treatment for patients with atrial fibrillation at discharge | 1 year
  The rate of patients with cerebral infarction complicated with atrial fibrillation who received anticoagulants (e.g., heparin, low molecular heparin, warfarin, new oral anticoagulants) at discharge in the total number of patients with cerebral infarction complicated with atrial fibrillation treated in hospital in the same period
Rate of blood vessel assessment within one week of hospitalization | 1 year
  The rate of patients with cerebral infarction hospitalized for 1 week who had completed the evaluation of the blood vessels in the neck and cranial (such as the ultrasound of the blood vessels in the neck or cranial, CT or MR angiography, or DSA) in the total number of cerebral infarction patients hospitalized in the same period

CONTACTS AND LOCATIONS:
Overall Officials: Zexin Chen, Principal Investigator — Tthe second affiliated hospital, school of medicine, Zhejiang University, China
Locations (1):
- Min Lou, Hangzhou, Zhejiang, China